CLINICAL TRIAL: NCT04226859
Title: Multicenter International Observational Study to Identify eGFR Trajectories and Their Determinants, and to Build a Multidimensional Prediction System to Predict the Probabilities of Belonging to eGFR Trajectories
Brief Title: Trajectories of Glomerular Filtration Rate and Progression to End Stage Renal Disease After Kidney Transplantation
Acronym: TRAJAKT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: TRAJAKT
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Kidney Transplant Failure; Kidney Function Issue
Keywords: Kidney Transplantation; Graft Survival; Glomerular Filtration Rate; Trajectories

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Kidney recipients aged over 18 and of all sexes recruited from 2000 in European and North American centers, who have eGFR follow-up and data from protocol and for cause biopsies available for allograft survival assessment; Randomized controlled trials conducted over the past 20 years with available data on protocol biopsy within the first year and follow up clinical, biological and histological data.

SUMMARY:
The gold standard for characterizing chronic kidney disease (CKD) is the glomerular filtration rate (GFR), which is commonly estimated in both native and transplanted kidneys for patient monitoring and therapeutic management and ultimately guides decision-making about whether a patient needs renal replacement therapy. In particular, the National Kidney Foundation has defined CKD stages according to estimated GFR (eGFR) values and in several studies, the eGFR slope or change has been found to be strongly associated with end stage renal disease (ESRD).

However, little is known about the heterogeneity of eGFR evolution in time - i.e. eGFR trajectories - and the related progression to ESRD and death. To date, no studies have investigated eGFR trajectories in diversified cohorts and populations worldwide, although this approach could provide a better understanding of CKD evolution and hence improve risk stratification. In addition, determinants of eGFR trajectories remain poorly described.

An unsupervised approach could allow examining eGFR trajectories over time and could lead to the identification of patient groups according to the probability of the progression of their kidney disease.

Therefore, this study aims:

1. To identify the long-term eGFR trajectories after kidney transplantation using latent class mixed models;
2. To identify the clinical, immunological, histological and functional determinants of the eGFR trajectories using multinomial regressions;
3. To investigate the associations of the eGFR trajectories with the progression to ESRD and death.

Based on the results, the investigators will provide an easily accessible tool to calculate personalized probabilities of belonging to eGFR trajectories after kidney transplantation, by using datasets from prospective cohorts and post hoc analysis of randomized control trial datasets.

DETAILED DESCRIPTION:
Background

Chronic kidney disease (CKD) now affects 850 million individuals worldwide, exceeding the global prevalence of diabetes, cancer and HIV/AIDS. In addition, end-stage renal disease affects 7.4 million individuals and mortality rate for individuals burdened by kidney disease is now estimated at 5 to 10 million individuals each year. Therefore, developing better diagnostic and treatment approaches for the kidney disease epidemic is a global priority, as leading professional societies and health agencies have emphasized (the US Food & Drug Administration, the National Kidney Foundation, the European Medicines Agency, the European Society of Organ Transplantation, the American Society for Transplantation and the American Society of Transplant Surgeons).

However, current approaches for investigating the relationship between eGFR course and outcomes such as ESRD and mortality have been limited by registries with an overall lack on granular data, including infrequent eGFR measurements for a single patient and convenience clinical samples. An unsupervised longitudinal approach to determine patient eGFR evolution may bring an original perspective to the traditional clinical interpretation of kidney function based on limited eGFR measurements, short-term follow-up, and standard statistical approach.

Main Outcome(s) and Measure(s)

* eGFR trajectories
* Determinants of eGFR trajectories
* Associations of eGFR trajectories with ESRD and death
* Prediction system that will provide the personalized probabilities of belonging to eGFR trajectories

ELIGIBILITY:
Inclusion Criteria:

* Kidney recipients transplanted after 2000
* Kidney recipients over 18 years of age
* Kidney recipients with at least two eGFR measurements after transplantation

Exclusion Criteria:

* Combined transplantation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Kidney recipients aged over 18 and of all sexes recruited from 2000 in European and North American centers, who have eGFR repeated measurements, data from protocol and for cause biopsies, as well as immunological, clinical, functional parameters and survival data for allograft and patient survival assessment. Additional kidney recipients from RCTs with longitudinal data including baseline and follow-up clinical, functional, immunological and histological data.
Sampling Method: Non-Probability Sample
Enrollment: 14000 (Estimated)
Dates: Start 2000-01 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
eGFR trajectories | Up to 10 years after kidney transplantation
  eGFR trajectories probabilities, calculated from a prediction system (based on clinical, histological, immunological, and functional factors) assessed at 1-year post transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, Professor, Principal Investigator — Paris Translational Research Center for Organ Transplantation
Locations (15):
- United States (5):
  - Department of Medicine, Division of Nephrology, Comprehensive Transplant Center, Cedars Sinai Medical Center, Los Angeles, California
  - Department of Surgery, Johns Hopkins University School of Medicine, Baltimore, Maryland
  - William J. von Liebig Center for Transplantation and Clinical Regeneration, Mayo Clinic, Rochester, Minnesota
  - Albert Einstein College of Medicine, Renal Division Montefiore Medical Center, Kidney Transplantation Program, New York, New York
  - Virginia Commonwealth University School of Medicine, Richmond, Virginia
- Department of Nephrology and Renal Transplantation, University Hospitals Leuven, Leuven, Belgium
- Department of Nephrology, Arterial Hypertension, Dialysis and Transplantation, University Hospital Centre Zagreb, School od Medicine University of Zagreb, Zagreb, Croatia
- France (8):
  - Department of Nephrology, Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Nephrology Dialysis Transplantation Department, University of Lorraine, Centre Hospitalier Universitaire de Nancy, Nancy
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Kidney Transplant Department, Saint-Louis Hospital, Assistance Publique - Hôpitaux de Paris, Paris
  - Kidney Transplant Department, Necker Hospital, Assistance Publique - Hôpitaux de Paris, Paris
  - Department of Transplantation, Nephrology and Clinical Immunology, Hôpital Foch, Suresnes
  - Department of Nephrology and Organ Transplantation, Centre Hospitalier Universitaire Rangueil, Toulouse
  - Bretonneau Hospital, Nephrology and Immunology Department, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Paris Transplant Group Website — https://www.paristransplantgroup.org